CLINICAL TRIAL: NCT02989675
Title: SugarFACT - Sugar Requirements For African Children Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Helena Hildenwall (Other)
Collaborators: Kamuzu University of Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Helena Hildenwall, MD, PhD, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.01/16/1852
Record Dates: First submitted 2016-12-05; First posted 2016-12-12 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Hypoglycemia Non Diabetics; Emergencies; Pediatric ALL; Critical Illness
Keywords: pediatric; critical illness; Malawi
MeSH Terms: conditions — Emergencies; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Critical Illness | interventions — Glucose

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dextrose (Experimental): Children in the intervention group will immediately receive intravenous 5ml/kg 10% dextrose, Dextrose administration will continue as a maintenance infusion of intravenous 10% dextrose for 24 hours at standard maintenance rates. Capillary blood glucose monitoring will be repeated at 30 minute intervals with repeated equivalent bolus doses given until levels reach ≥5.0mmol/l. All children will be kept in the emergency department for a minimum of 60 minutes and have their vital signs checked at discharge from the emergency room to the ward.
  Interventions: Drug: 10% dextrose
- Control (No Intervention): Usual care - the care that is currently provided in the hospital - will be provided. All children in the control group will be kept in the emergency department for a minimum of 60 minutes and have their vital signs checked at discharge from the emergency room to the ward.

INTERVENTIONS:
Drug: 10% dextrose — Bolus of 10% dextrose 5mls/kg
  Arms: Dextrose

SUMMARY:
The purpose of this study is to evaluate the impact of dextrose administration in severely sick children admitted to hospital with low-glycaemia.

The problem: Mortality in children remains high in sub-Saharan African hospitals. While antimalarial drugs, antibiotics and other definitive treatments are well understood, the role of emergency care with supportive therapies such as maintaining normal glucose and electrolyte balances, has been given limited attention. Hypoglycaemia is common in children admitted to hospital in low-income settings. The current definition of hypoglycaemia is a blood glucose level of less than 2.5mmol/l. Outcomes for these children are poor, with a mortality rate of up to 42%. An increased mortality has also been reported among acutely ill children with low-glycaemia, defined as a blood glucose level of 2.5-5.0mmol/l. The reason for increased mortality rates is not fully understood.

Study objective: To determine the impact on mortality of a raised treatment cut-off level for paediatric hypoglycaemia, from 2.5mmol/l to 5.0mmol/l.

Methodology: Severely ill children admitted to two central Malawian hospitals; Queen Elisabeth Central Hospital, Blantyre and Zomba Central Hospital, with low-glycaemia (2.5-5.0mmol/l) will be randomised into intervention or control groups. The intervention group will be treated with an intravenous bolus of 10% dextrose 5ml/kg followed by a dextrose infusion in addition to standard care while the control group will receive standard care only. Children will be followed until discharge from hospital or death. Primary end-point is in-hospital mortality.

DETAILED DESCRIPTION:
Enrolment started at Queen Elisabeth Central Hospital on Dec 5th 2016. Due to a slow enrolment rate a second site at Zomba Central Hospital has been opened to start enrolment on October 17th, 2017 in order for the project to be completed in December 2019.

ELIGIBILITY:
Inclusion Criteria:

* Age between one month to 5 years (5 to 12 years for outcome measure no 3)
* Parent/carer willing and able to give consent
* Presence of one or several emergency signs (as defined in WHO pocket book of hospital care for children)

  * Obstructed or absent breathing
  * Central cyanosis
  * Severe respiratory distress
  * Shock/impaired perfusion
  * Coma/reduced consciousness
  * Convulsions
  * Severe dehydration
* Clinical concern that the child is in an emergency state
* Blood glucose 2.5-5.0mmol/l at arrival to the emergency department (3.0-5.0mmol/l for severely malnourished children). For outcome measure no 4 children with <2.5 mmol/l on arrival who then have 2.5-5.0 mmol/l on the repeat test 30 minutes later are also included

Exclusion Criteria:

* Children with a known diagnosis of diabetes
* Refusal to participate by the child or guardians

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 410 (Actual)
Dates: Start 2016-12; Primary Completion 2019-01-22 (Actual); Study Completion 2019-01-22 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality in children 1 month to 5 years old | Up to 12 months
  From date of randomization until the date of discharge from hospital or date of in-hospital death, whichever came first, assessed up to 12 months

SECONDARY OUTCOMES:
24 hours mortality in children 1 month to 5 years old | 24 hours after admission
  Mortality within the first 24 hrs after admission

OTHER OUTCOMES:
In-hospital mortality in children 5-12 years old | Up to 12 months
  From date of randomization until the date of discharge from hospital or date of in-hospital death, whichever came first, assessed up to 12 months
In hospital mortality in children with initial hypoglycaemia (blood glucose <2.5mmol/l) and low glycemia after first dextrose bolus | Up to 12 months
  From date of randomization until the date of discharge from hospital or date of in-hospital death, whichever came first, assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Helena Hildenwall, MD, PhD, Principal Investigator — Karolinska Institutet; Tim Baker, MD, PhD, Principal Investigator — Karolinska Institutet; Queen Dube, MD, PhD, Principal Investigator — College of Medicine, Malawi; Josephine Langton, MD, Principal Investigator — College of Medicine, Malawi
Locations (2):
- Malawi (2):
  - Queen Elisabeth Central Hospital, Blantyre
  - Zomba Central Hospital, Zomba

REFERENCES:
- [Derived] Baker T, Ngwalangwa F, Masanjala H, Dube Q, Langton J, Marrone G, Hildenwall H. Effect on mortality of increasing the cutoff blood glucose concentration for initiating hypoglycaemia treatment in severely sick children aged 1 month to 5 years in Malawi (SugarFACT): a pragmatic, randomised controlled trial. Lancet Glob Health. 2020 Dec;8(12):e1546-e1554. doi: 10.1016/S2214-109X(20)30388-0. Epub 2020 Oct 8. PMID 33038950
- [Derived] Baker T, Dube Q, Langton J, Hildenwall H. Mortality impact of an increased blood glucose cut-off level for hypoglycaemia treatment in severely sick children in Malawi (SugarFACT trial): study protocol for a randomised controlled trial. Trials. 2018 Jan 11;19(1):33. doi: 10.1186/s13063-017-2411-8. PMID 29325595